CLINICAL TRIAL: NCT02515604
Title: Comparison of Single and Repeated Dose of Vaginal Misoprostol for the Treatment of Early Pregnancy Failure - a Randomized Clinical Trial
Brief Title: Comparison of Single and Repeated Dose of Vaginal Misoprostol for the Treatment of Early Pregnancy Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Yossi Mizrachi, MD, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0104-15-WOMC
Record Dates: First submitted 2015-08-02; First posted 2015-08-05 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Abortion, Missed
MeSH Terms: conditions — Abortion, Missed | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose group (Active Comparator)
  Interventions: Drug: Misoprostol
- Repeated dose group (Active Comparator)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol
  Other Names: Cytotec

SUMMARY:
A randomised controlled trial assessing the efficacy of single versus repeated dose of vaginal misoprostol for the treatment of early pregnancy failure.

ELIGIBILITY:
Inclusion Criteria:

* Women with early pregnancy failure, defined as missed abortion or blighted ovum, seeking medical treatment with misoprostol.
* Age equal or greater than 18 years
* Gestational age less than 12 complete weeks.

Exclusion Criteria:

* Complete, incomplete, inevitable, or septic abortion.
* Hemodynamically unstable patients.
* Misoprostol sensitivity or contraindication.
* Multifetal pregnancies.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Complete abortion (Endometrial thickness of less than 15 mm, as assessed by trans-vaginal ultrasound.) | Day 8 from first misoprostol dose
  Endometrial thickness of less than 15 mm, as assessed by trans-vaginal ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Yossi Mizrachi, MD, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson Medical Center, Holon, Israel

REFERENCES:
- [Derived] Mizrachi Y, Dekalo A, Gluck O, Miremberg H, Dafna L, Feldstein O, Weiner E, Bar J, Sagiv R. Single versus repeat doses of misoprostol for treatment of early pregnancy loss-a randomized clinical trial. Hum Reprod. 2017 Jun 1;32(6):1202-1207. doi: 10.1093/humrep/dex074. PMID 28402415